CLINICAL TRIAL: NCT00290485
Title: A Phase II Study on Preoperative Administration of Gleevec in Patients With Initially Non-Resectable Gastrointestinal Stromal Tumor
Brief Title: Gleevec Administered Preoperatively to Reduce Gastrointestinal Stromal Tumor (GIST)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Collaborators: Hippocrate Research & Development (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Q-CTG-01-V7.0-A1; NCT00363103 (obsolete NCT alias)
Record Dates: First submitted 2006-02-09; First posted 2006-02-13 (Estimated); Last update posted 2006-04-07 (Estimated); Status verified 2006-04

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: non-resectable tumor; high-risk tumor; metastasis; Response Evaluation Criteria in Solid Tumors (RECIST); Gleevec; Imatinib mesylate
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Neoplasm Metastasis | interventions — Imatinib Mesylate

INTERVENTIONS:
Drug: Imatinib mesylate

SUMMARY:
The aim of this study is to demonstrate that the use of Gleevec in initially non-resectable gastrointestinal stromal tumors can lead to allow complete resection in 20% of cases.

DETAILED DESCRIPTION:
Gastrointestinal stromal tumor (GIST) is a specific, immunohistochemically KIT+ mesenchymal neoplasm of the gastrointestinal tract. The identification of KIT+ tumor has become more important after introduction of target treatment with KIT tyrosine kinase inhibitor Imatinib mesylate (Gleevec). Despite this progress, GIST patients presenting a tumor larger than 5 cm have a 10 year survival between 10% and 30%. Indeed, the risk of microscopic spreading of the tumor during surgery is very high since intra-abdominal organs are in close relation to each others. To improve survival, it seemed logical to use preoperative Gleevec to reduce tumor size and improve efficacy of the surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* GIST patient considered initially non-resectable as defined by one of the following:

  1. when the surgical team considers that the risk of incomplete resection (R1 or R2) of a GIST is higher than 20%
  2. when the resection of a GIST necessitates a highly morbid procedure
  3. when a GIST is attached to 3 or more major intra-abdominal structures or to a major intra-abdominal blood vessel
  4. when GIST is considered at very high risk of recurrence. This is the case when it is a recurrence or when the tumor is in very close contact with a structure that cannot be resected by surgery or when the patient has metastasis.
* Outpatient is 18 years old or more
* ECOG performance status 0, 1 or 2
* Immunohistochemical confirmation of KIT overexpression must exist at the study entry
* Measurable disease on CT-Scan or MRI (ultrasound and/or operative finding are not acceptable) and response to RECIST criteria
* Have a life expectancy of at least 6 months
* Be willing and able to comply with the protocol (and surgery if required) for the duration of the study
* Give written informed consent prior to study-specific screening procedure, with the understanding that the patient has the right to withdraw from the study at any time without prejudice

Exclusion Criteria:

* received Imatinib in the past
* received a full course of radiotherapy within 3 months of inclusion in the study. A short course of radiotherapy to control bleeding is allowed.
* received systemic chemotherapy within 4 weeks of inclusion in the study
* received steroids for less than 4 weeks of inclusion in the study
* pregnant or lactating women
* women of childbearing potential with either a positive or no pregnancy test at baseline. Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential.
* sexually active males or females (of childbearing potential) unwilling to practice contraception during the study
* history of other malignancy within the past 5 years, except cured basal cell carcinoma of skin and cured carcinoma in-situ of uterine cervix
* clinical or other evidence of CNS metastases
* myocardial infarction within the last 3 months
* any medical condition that contraindicates potential surgery
* lack of physical integrity of the upper gastrointestinal tract, malabsorption syndrome or inability to take oral medication
* any serious uncontrolled concomitant disease
* any of the following laboratory values:

  1. absolute neutrophil count < 1.5 E+09/L
  2. platelet count < 80000 E+09/L
  3. AST or ALT higher than 2 X normal
* major surgery within 4 weeks prior to start of study treatment, or lack of complete recovery from effects of major surgery
* patients with known or suspected hypersensitivity to one of the Gleevec components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2005-08

PRIMARY OUTCOMES:
Patient response rate according to RECIST criteria

SECONDARY OUTCOMES:
Clinical response to treatment
Radiological response to treatment
Pathological response to treatment
Compare clinical with pathological response
Evaluate the impact of Gleevec on surgical morbidity
Evaluate disease-free survival
Evaluate overall survival
Evaluate whether the response rate can predict survival

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Dubé, MD, Study Chair — Maisonneuve-Rosemont Hospital
Locations (1):
- Maisonneuve-Rosemont Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] Kitamura Y, Hirota S, Nishida T. Gastrointestinal stromal tumors (GIST): a model for molecule-based diagnosis and treatment of solid tumors. Cancer Sci. 2003 Apr;94(4):315-20. doi: 10.1111/j.1349-7006.2003.tb01439.x. PMID 12824897
- [Background] Judson I. Gastrointestinal stromal tumours (GIST): biology and treatment. Ann Oncol. 2002;13 Suppl 4:287-9. doi: 10.1093/annonc/mdf672. No abstract available. PMID 12401703
- [Background] Greenson JK. Gastrointestinal stromal tumors and other mesenchymal lesions of the gut. Mod Pathol. 2003 Apr;16(4):366-75. doi: 10.1097/01.MP.0000062860.60390.C7. PMID 12692202
- [Background] Rosai J. GIST: an update. Int J Surg Pathol. 2003 Jul;11(3):177-86. doi: 10.1177/106689690301100304. No abstract available. PMID 12894349
- [Background] Bono P, Krause A, von Mehren M, Heinrich MC, Blanke CD, Dimitrijevic S, Demetri GD, Joensuu H. Serum KIT and KIT ligand levels in patients with gastrointestinal stromal tumors treated with imatinib. Blood. 2004 Apr 15;103(8):2929-35. doi: 10.1182/blood-2003-10-3443. Epub 2004 Jan 8. PMID 15070666
- [Background] Schirru A, Cavaliere D, Cosce U, Scarimbolo M, Griseri G, Caristo I, Bianchi M, Ingravaglieri E, Aiello D, Venturino E. [Surgical treatment of gastrointestinal stromal tumors: personal cases]. Tumori. 2003 Jul-Aug;89(4 Suppl):141-2. Italian. PMID 12903574
- [Background] Liberati G, Lucchetta MC, Petraccia L, Nocchi S, Rosentzwig R, De Matteis A, Grassi M. [Meta-analytical study of gastrointestinal stromal tumors (GIST)]. Clin Ter. 2003 Mar-Apr;154(2):85-91. Italian. PMID 12856366
- [Background] Kanda T, Ohashi M, Makino S, Kaneko K, Matsuki A, Nakagawa S, Hatakeyama K. A successful case of oral molecularly targeted therapy with imatinib for peritoneal metastasis of a gastrointestinal stromal tumor. Int J Clin Oncol. 2003 Jun;8(3):180-3. doi: 10.1007/s10147-003-0321-0. PMID 12851843
- [Background] Miettinen M, Lasota J. Gastrointestinal stromal tumors (GISTs): definition, occurrence, pathology, differential diagnosis and molecular genetics. Pol J Pathol. 2003;54(1):3-24. PMID 12817876
- [Background] DeMatteo RP. The GIST of targeted cancer therapy: a tumor (gastrointestinal stromal tumor), a mutated gene (c-kit), and a molecular inhibitor (STI571). Ann Surg Oncol. 2002 Nov;9(9):831-9. doi: 10.1007/BF02557518. PMID 12417503
- [Background] Tuveson DA, Willis NA, Jacks T, Griffin JD, Singer S, Fletcher CD, Fletcher JA, Demetri GD. STI571 inactivation of the gastrointestinal stromal tumor c-KIT oncoprotein: biological and clinical implications. Oncogene. 2001 Aug 16;20(36):5054-8. doi: 10.1038/sj.onc.1204704. PMID 11526490
- [Background] Blanke CD, Eisenberg BL, Heinrich MC. Gastrointestinal stromal tumors. Curr Treat Options Oncol. 2001 Dec;2(6):485-91. doi: 10.1007/s11864-001-0070-0. PMID 12057094
- [Background] Yan H, Marchettini P, Acherman YI, Gething SA, Brun E, Sugarbaker PH. Prognostic assessment of gastrointestinal stromal tumor. Am J Clin Oncol. 2003 Jun;26(3):221-8. doi: 10.1097/01.COC.0000018296.45892.CE. PMID 12796588
- [Background] Noguchi T, Sato T, Takeno S, Uchida Y, Kashima K, Yokoyama S, Muller W. Biological analysis of gastrointestinal stromal tumors. Oncol Rep. 2002 Nov-Dec;9(6):1277-82. PMID 12375034
- [Background] Kovac D, Petrovecki M, Jasic M, Dobi-Babic R, Ivanis N, Rubinic M, Krizanac S, Jonjic N, Rizzardi C, Melato M. Prognostic factors of gastrointestinal stromal tumors. Anticancer Res. 2002 May-Jun;22(3):1913-7. PMID 12168893
- [Background] Connolly EM, Gaffney E, Reynolds JV. Gastrointestinal stromal tumours. Br J Surg. 2003 Oct;90(10):1178-86. doi: 10.1002/bjs.4352. PMID 14515284
- [Background] Crosby JA, Catton CN, Davis A, Couture J, O'Sullivan B, Kandel R, Swallow CJ. Malignant gastrointestinal stromal tumors of the small intestine: a review of 50 cases from a prospective database. Ann Surg Oncol. 2001 Jan-Feb;8(1):50-9. doi: 10.1007/s10434-001-0050-4. PMID 11206225
- [Background] Joensuu H. Treatment of inoperable gastrointestinal stromal tumor (GIST) with Imatinib (Glivec, Gleevec). Med Klin (Munich). 2002 Jan 15;97 Suppl 1:28-30. PMID 11831069
- [Background] Rajput A, Kraybill WG. Clinical trials and soft tissue sarcomas. Surg Oncol Clin N Am. 2003 Apr;12(2):485-97. doi: 10.1016/s1055-3207(03)00002-4. PMID 12916465
- [Background] Patel SR. Systemic therapy for advanced soft-tissue sarcomas. Curr Oncol Rep. 2002 Jul;4(4):299-304. doi: 10.1007/s11912-002-0005-3. PMID 12044239
- [Background] Eisenberg BL. Imatinib mesylate: a molecularly targeted therapy for gastrointestinal stromal tumors. Oncology (Williston Park). 2003 Nov;17(11):1615-20; discussion 1620, 1623, 1626 passim. PMID 14682111
- [Background] Rossi CR, Mocellin S, Mencarelli R, Foletto M, Pilati P, Nitti D, Lise M. Gastrointestinal stromal tumors: from a surgical to a molecular approach. Int J Cancer. 2003 Nov 1;107(2):171-6. doi: 10.1002/ijc.11374. PMID 12949790
- [Background] Radford IR. Imatinib. Novartis. Curr Opin Investig Drugs. 2002 Mar;3(3):492-9. PMID 12054102
- [Background] Frolov A, Chahwan S, Ochs M, Arnoletti JP, Pan ZZ, Favorova O, Fletcher J, von Mehren M, Eisenberg B, Godwin AK. Response markers and the molecular mechanisms of action of Gleevec in gastrointestinal stromal tumors. Mol Cancer Ther. 2003 Aug;2(8):699-709. PMID 12939459
- [Background] Demetri GD, von Mehren M, Blanke CD, Van den Abbeele AD, Eisenberg B, Roberts PJ, Heinrich MC, Tuveson DA, Singer S, Janicek M, Fletcher JA, Silverman SG, Silberman SL, Capdeville R, Kiese B, Peng B, Dimitrijevic S, Druker BJ, Corless C, Fletcher CD, Joensuu H. Efficacy and safety of imatinib mesylate in advanced gastrointestinal stromal tumors. N Engl J Med. 2002 Aug 15;347(7):472-80. doi: 10.1056/NEJMoa020461. PMID 12181401
- [Background] Bumming P, Andersson J, Meis-Kindblom JM, Klingenstierna H, Engstrom K, Stierner U, Wangberg B, Jansson S, Ahlman H, Kindblom LG, Nilsson B. Neoadjuvant, adjuvant and palliative treatment of gastrointestinal stromal tumours (GIST) with imatinib: a centre-based study of 17 patients. Br J Cancer. 2003 Aug 4;89(3):460-4. doi: 10.1038/sj.bjc.6600965. PMID 12888812